CLINICAL TRIAL: NCT01278823
Title: Effect of Bariatric Surgery on Mechanisms of Type 2 Diabetes
Acronym: STAMPEDEII
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Cleveland Clinic (Other)
Responsible Party: Principal Investigator, Philip Schauer, MD, The Cleveland Clinic
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1R01DK089547 (NIH)
Record Dates: First submitted 2011-01-17; First posted 2011-01-19 (Estimated); Last update posted 2019-07-11 (Actual); Status verified 2019-07

CONDITIONS: Obesity; Type 2 Diabetes
Keywords: obesity; type 2 diabetes
MeSH Terms: conditions — Obesity; Diabetes Mellitus, Type 2 | interventions — Bariatric Surgery; Practice Management, Medical; Exercise; Self-Help Groups

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- surgery (Experimental): Surgery: laparoscopic roux en y gastric bypass operation
  Interventions: Procedure: laparoscopic roux en y gastric bypass operation
- Medical treatment (Active Comparator): Medical Treatment: Comprehensive medical management of diabetes including medications, diet intervention, lifestyle modification, exercise regimen
  Interventions: Other: medical management

INTERVENTIONS:
Procedure: laparoscopic roux en y gastric bypass operation — roux en y gastric bypass operation
  Other Names: bariatric surgery
  Arms: surgery
Other: medical management — latest type 2 diabetes medications, lifestyle/behavior modification and dietary regimen
  Other Names: meal replacement; exercise; group support
  Arms: Medical treatment

SUMMARY:
The purpose of this study is to determine the effects of bariatric surgery on blood sugar control and underlying mechanisms that contribute to type 2 diabetes in men and women with a BMI between 27 and 42. Sixty subjects will be randomized to either undergo the roux-en-y gastric bypass operation or intensive medical, dietary and exercise management.

DETAILED DESCRIPTION:
Obesity and type 2 diabetes mellitus (T2DM) are two of the greatest public health problems of the 21st century. Lifestyle changes and pharmacotherapy, which are mainstay treatments for T2DM have had limited success. More intensive lifestyle weight management such as in the Look AHEAD trial reported an 8.6% weight loss after 1 year, while the Diabetes Prevention Program reported a 7% weight loss after 2 years, and a 58% decrease in the risk of developing T2DM. In contrast,we have observed a 31% weight loss together with 83% remission of T2DM in severely obese patients after Roux-en-Y gastric bypass (RYGB) surgery. However, direct evidence of the glycemic benefits of bariatric surgery from randomized control trials is lacking; there is no clear consensus that RYGB surgery is a good treatment option for moderately obese T2DM patients; and the mechanisms responsible for reversing T2DM after surgery remain unclear but may involve pancreatic insulin secretion and skeletal muscle and hepatic insulin resistance.

The objective of this application is to evaluate the effects of RYGB surgery on glycemic control and underlying mechanisms that contribute to T2DM in obese subjects (BMI: 30-40 kg/m2). Our central hypothesis is that RYGB surgery will reduce hyperglycemia via reversal of beta-cell dysfunction and decrease hepatic and peripheral insulin resistance. The approach requires a 12-month randomized controlled trial. The rationale is based on data showing that RYGB lowers fasting and postprandial glucose, and increases the GLP-1 response to a meal. However, the therapeutic efficacy of RYGB surgery in obesity-related T2DM needs to be demonstrated in a randomized trial.

ELIGIBILITY:
Inclusion Criteria:

* candidate for general surgery
* 18 to 60 years old
* BMI 27-43
* type 2 diabetes
* willing to participate in either study arm
* understand and comply with requirements of each arm
* not pregnant
* willing to use reliable birth control for duration of study

Exclusion Criteria:

* prior bariatric surgery of any type
* prior complex abdominal surgery
* abdominal, thoracic, pelvic, obstetrical surgery within last 6 months
* significant cardiovascular disease
* kidney disease with a creatinine greater than or equal to 1.8 mg/dl
* chronic liver disease except for NAFLD/NASH
* celiac, malabsorptive, inflammatory bowel disorders
* psychiatric disorders requiring 3 or more medications
* pregnancy
* cancer except squamous or basal cell skin cancer or cancer in remission
* anticoagulation therapy that can't be stopped for surgery
* clotting disorders
* severe pulmonary disease

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 18 (Actual)
Dates: Start 2011-01; Primary Completion 2017-02-15 (Actual); Study Completion 2017-02-15 (Actual)

PRIMARY OUTCOMES:
Test the effect of gastric bypass surgery on glycemic control in obese type 2 DM patients | 12 months
  The working hypothesis for this aim is that significantly more obese T2DM patients who undergo RYGB surgery will achieve glycemic control based on a primary endpoint of an HbA1c ≤ 6.5% at 12 months, than patients managed by intensive medical therapy.

SECONDARY OUTCOMES:
Determine the effects of gastric bypass surgery on pancreatic beta cell function and incretin hormone secretion in obese type 2 dm patients | 12 months
  The working hypothesis for this aim is that a primary physiological link between obesity and T2DM is specific to beta-cell dysfunction; RYGB will reverse beta-cell dysfunction by increasing postprandial incretin secretion.

CONTACTS AND LOCATIONS:
Overall Officials: John Kirwan, PhD, Principal Investigator — The Cleveland Clinic
Locations (1):
- Cleveland Clinic Bariatric and Metabolic Institute, Department of Pathobiology, Cleveland, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kirwan JP, Axelrod CL, Kullman EL, Malin SK, Dantas WS, Pergola K, Del Rincon JP, Brethauer SA, Kashyap SR, Schauer PR. Foregut Exclusion Enhances Incretin and Insulin Secretion After Roux-en-Y Gastric Bypass in Adults With Type 2 Diabetes. J Clin Endocrinol Metab. 2021 Sep 27;106(10):e4192-e4201. doi: 10.1210/clinem/dgab255. PMID 33870426
- See also: Cleveland Clinic Bariatric and Metabolic Institute web site — https://weightloss.clevelandclinic.org